CLINICAL TRIAL: NCT00414921
Title: Preschool Supplement to Clonidine in ADHD (Kiddie-CAT)
Acronym: kiddie-CAT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Cincinnati (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Floyd R. Sallee, M.D., Ph.D., Professor, University of Cincinnati School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R01NS39087_kiddie-CAT; R01NS039087 (NIH)
Record Dates: First submitted 2006-12-21; First posted 2006-12-22 (Estimated); Last update posted 2009-05-21 (Estimated); Status verified 2007-12

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: Attention deficit hyperactivity disorder; ADHD; clonidine; methylphenidate; MPH
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Clonidine; Methylphenidate; 5,10-dihydro-5-methylphenazine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Active Comparator): clonidine
  Interventions: Drug: clonidine
- 2 (Active Comparator): methylphenidate
  Interventions: Drug: methylphenidate
- 3 (Active Comparator): methylphenidate and clonidine
  Interventions: Drug: clonidine; Drug: methylphenidate
- 4 (Placebo Comparator)
  Interventions: Other: placebo

INTERVENTIONS:
Drug: clonidine — Clonidine is FDA-approved for the treatment of hypertension in adults
  Arms: 1; 3
Drug: methylphenidate — Methylphenidate is known to safely and effectively treat many ADHD symptoms.
  Other Names: MPH
  Arms: 2; 3
Other: placebo — inactive substance
  Arms: 4

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of two medications--clonidine and methylphenidate--alone or in combination to treat attention deficit hyperactivity disorder in children ages 4 through 6.

DETAILED DESCRIPTION:
Attention deficit hyperactivity disorder (ADHD) is a disease characterized by one or more symptoms of hyperactivity, impulsivity, or inattention that interfere with school, home, work, or social settings. ADHD does not have clear physical signs that can be seen in an x-ray or a lab test. The disorder only can be identified by looking for certain behaviors, which vary from person to person.

This trial will compare the benefits and side effects of two medications--clonidine and methylphenidate (MPH)--used alone or in combination to treat ADHD in children. MPH is approved by the Food and Drug Administration (FDA) for the treatment of ADHD symptoms in children, and clonidine is FDA-approved for the treatment of hypertension in adults. Stimulant medications such as MPH are known to safely and effectively treat many ADHD symptoms. Such medicines, however, do not cure the condition or improve all ADHD symptoms, and the long-term effectiveness of these medications is not well-known.

In this study, participants will be randomly selected to receive one of four treatments: 1) clonidine; 2) MPH; 3) clonidine and MPH; or 4) a placebo (an inactive substance). Participation in the study is about 16 weeks, and includes a baseline screening and 5 evaluation visits to assess attention, hyperactivity, overall improvement and general functioning, medication side effects, blood pressure, pulse, and weight.

ELIGIBILITY:
Inclusion Criteria:

* Child with ADHD
* Child ages 4 through 6
* Child attending a structured preschool or daycare

Exclusion Criteria:

* Presence of a tic disorder of any kind or a known active heart disease for which it would be unsafe to use the study drugs
* Presence of pervasive developmental disorder, autism, mental retardation, or serious psychiatric illness
* Child not attending a structured preschool or daycare

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2003-09; Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
change in score on the Conners Abbreviated Symptom Questionnaire for Teachers (ASQ-T) | at 16 weeks

SECONDARY OUTCOMES:
the ASQ-Parent (ASQ-P) and Child Global Assessment Scales (C-GAS). Adverse events were monitored using AE logs, the Pittsburgh Side Effects Rating Scale, vital signs and electrocardiograms. | at 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Floyd Randy Sallee, MD/PhD, Principal Investigator — University of Cincinnati; Oscar Bukstein, MD, Principal Investigator — Western Psychiatric Institute and Clinic; Donna Palumbo, PhD, Principal Investigator — University of Rochester; William Pelham, PhD, Principal Investigator — SUNY Buffalo
Locations (3):
- United States (3):
  - University of Rochester Medical Center, Department of Neurology, 919 Westfall Road, Building C, Rochester, New York
  - University of Cincinnati, Department of Psychiatry, 231 Albert Sabin Way, M: 0559, Cincinnati, Ohio
  - Western Psychiatric Institute and Clinic, ADD Program, 3811 Ohara Street, Pittsburgh, Pennsylvania